CLINICAL TRIAL: NCT00278954
Title: A Phase III, Multicenter, Open-Label Study To Evaluate The Efficacy, Safety, and Pharmacokinetics of Gammaplex® in Primary Immunodeficiency Diseases
Brief Title: Efficacy, Safety and Pharmacokinetics of Gammaplex in Primary Immunodeficiency Diseases.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMX01
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Primary Immunodeficiency; Common Variable Hypogammaglobulinemia; X-linked Hypogammaglobulinemia; Hypogammaglobulinemia; Immunodeficiency With Hyper-IgM; Wiskott-Aldrich Syndrome
Keywords: Primary Antibody Deficiency; Common variable hypogammaglobulinemia; X-linked hypogammaglobulinemia; Hypogammaglobulinemia; Immunodeficiency with hyper-IgM; Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Hypogammaglobulinemia, X-Linked; Agammaglobulinemia; Hyper-IgM Immunodeficiency Syndrome; Wiskott-Aldrich Syndrome | interventions — gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gammaplex (Other): Gammaplex
  Interventions: Biological: Gammaplex (Intravenous immunoglobulin)

INTERVENTIONS:
Biological: Gammaplex (Intravenous immunoglobulin) — GAMMAPLEX 5g/100 mL, dose is 300-800 mg/kg/infusion every 21 or 28 days, intravenously for 12 months.

SUMMARY:
The main objective of this study is to see if GAMMAPLEX is efficacious with respect to Food and Drug Administration (FDA) minimal requirements (no more than 1 serious, acute, bacterial infection per subject per year) in subjects with Primary Immunodeficiency Diseases (PID). The secondary objectives are to assess the safety and tolerability of GAMMAPLEX and to determine if GAMMAPLEX has a pharmacokinetic (PK) profile comparable with that of intact Immunoglobulin G (IgG) in subjects with PID.

DETAILED DESCRIPTION:
Primary Efficacy Variable The primary variable is the number of serious, acute, bacterial infections/subject/year, and it will be based on the total of all of the following events as defined by the FDA: bacterial Pneumonia, bacteremia/sepsis, osteomyelitis/septic arthritis, visceral abscess, and bacterial meningitis.

Secondary Efficacy Variables Secondary efficacy will be determined by using the following variables: number of days of work/school missed because of infection per subject year; number and days of hospitalizations because of infection per subject year; number of visits to physicians for acute problems and/or number of visits to hospital emergency rooms per subject year; other infections documented by fever or a positive result on a radiograph and/or culture; number of infectious episodes per subject per year; number of days on therapeutic antibiotics.These data will be entered into the subject diary, confirmed by the physician, and entered on the electronic-CRF (e-CRF).

Safety Variables. The variables used to assess safety will be the following: adverse events (AEs); vital signs; clinical laboratory tests and Direct Coombs' Test; transmission of viruses; physical examination.

Test product, dose/mode of administration, batch number(s): The GAMMAPLEX dose is 300-800 mg/kg/infusion (milligram per killgram per infusion) every 21 or 28 days, intravenously. At least 2 batches will be used in this study and no more than 1 batch in any given infusion.

Duration of treatment:

The total duration of treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject is 3 years of age or older, of either sex, belonging to any ethnic group, and above a minimum weight of 27.5 kg. This weight is based on the amount of blood required for testing. If subject is participating in the PK segment, the minimum weight required is 37 kg.

  2. The subject has a primary immunodeficiency disease, which has as a significant component of hypogammaglobulinemia and/or antibody deficiency (e.g. (exempli gratia / for example), common variable immunodeficiency, X-linked and autosomal forms of agammaglobulinemia, hyper-immunoglobulin M (hyper-IgM) syndrome, Wiskott-Aldrich Syndrome). Isolated deficiency of a single IgG subclass, or of specific antibodies without hypogammaglobulinemia per se, does not qualify for inclusion.

  3. The subject has been receiving licensed or investigational (Phase III or IIIb) immunoglobulin intravenous (IGIV) replacement therapy at a dose that has not changed by + 50% of the mean dose for at least 3 months before study entry and is between 300 and 800 mg/kg/infusion. The infusion interval must be between 21 and 28 days inclusive. The subject must have maintained a trough level at least 300 mg/dL (milligram per decilitre) above baseline serum IgG levels (defined as before initiation of any gamma globulin treatment for that subject). The trough level must be 600 mg/dL.

  4. Trough levels of IgG and dose of IGIV, treatment intervals, and the trade name of the IGIV treatments used for the last 2 consecutive routine (licensed or investigational product) must be documented for each subject before the first infusion in this study can be administered.

  5. If a subject is a female of child-bearing potential, she must have a negative result on an Human Chorionic Gonadotrophin (HCG)-based pregnancy test.

  6. If a subject is a female who is or becomes sexually active, she must practice contraception by using a method of proven reliability for the duration of the study.

  7. The subject is willing to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

  8. The subject has signed an informed consent form (if at least 18 years old) or the subject's parent or legal guardian has signed the informed consent form. If appropriate, the subject has signed a child assent form (See Section 12.3).

Exclusion Criteria:

* Subjects will be excluded if any of the following exclusion criteria are met:

  1. The subject has a history of any severe anaphylactic reaction to blood or any blood-derived product.
  2. The subject is known to be intolerant to any component of GAMMAPLEX, such as sorbitol (i.e.(id est / that is) , intolerance to fructose).
  3. The subject has selective immunoglobulin A (IgA) deficiency, history of reaction to products containing IgA, or has a history of antibodies to IgA.
  4. Subjects who have completed the study and subjects who have withdrawn cannot participate in the study for a second time.
  5. The subject is currently receiving, or has received, any investigational agent, other than an immune serum globulin (ISG) preparation that is being evaluated in a Phase III or IIIb study, within the prior 3 months.
  6. The subject has been exposed to blood or any blood product or derivative within the last 6 months, other than a commercially available IGIV or other forms of commercially available and licensed ISG or an ISG product that is in Phase III or IIIb studies.
  7. The subject is pregnant or is nursing.
  8. The subject is positive for any of the following at screening:

     * Serological test for Human immunodeficiency virus (HIV) 1&2, Hepatitis C virus (HCV), or Hepatitis B surface antigen (HBsAg)
     * Nucleic Acid test (NAT) for HCV
     * NAT for HIV
  9. The subject, at screening, has levels greater than 2.5 times the upper limit of normal as defined at the central laboratory of any of the following:

     * Alanine transaminase (ALT)
     * Aspartate transaminase (AST)
  10. The subject has a severe renal impairment (defined as serum creatinine greater than 2 times the upper limit of normal or Blood urea nitrogen (BUN) greater than 2.5 times the upper limit of normal for the range of the laboratory doing the analysis); the subject is on dialysis; the subject has a history of acute renal failure.
  11. The subject is known to abuse alcohol, opiates, psychotropic agents, or other chemicals or drugs, or has done so within the past 12 months.
  12. The subject has a history of deep vein thrombosis (DVT), or thrombotic complications of IGIV therapy.
  13. The subject suffers from any acute or chronic medical condition (e.g., renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing state) that, in the opinion of the investigator, may interfere with the conduct of the study.
  14. The subject has an acquired medical condition, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (Absolute neutrophil count (ANC) < 1000 x 109/L).
  15. The subject is receiving the following medication:

      * Immunosuppressive drugs
      * The subject is receiving the following medication: Steroids (long-term daily, >0.15 mg /kg/day of prednisone or prednisolone of equivalent dose of other corticosteroids) The requirement for burst or intermittent courses would not exclude the subject.
      * Immunomodulatory drugs
  16. The subject has non-controlled arterial hypertension (systolic blood pressure > 160 mmHg (millimeters of mercury) and/or diastolic blood pressure > 100 mmHg).
  17. The subject has anemia (hemoglobin < 10 g/dL) at screening.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Berger, MD, Principal Investigator — Rainbow Babies & Children's Hospital, Cleveland, Ohio
Locations (7):
- United States (7):
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Family Allergy and Asthma Center PC, Atlanta, Georgia
  - Rush University Medical Centre, University Consultants in Allergy & Immunology, Chicago, Illinois
  - Childrens Hospital at Buffalo, Allergy Division, Buffalo, New York
  - Allergy, Asthma & Immunology Clinic, P.A., Irving, Texas
  - UCLA Medical Centre, Irving, Texas
  - University of Washington School of Medicine, Dept. of Pediatrics, Seattle, Washington

REFERENCES:
- [Derived] Geng B, Clark K, Evangelista M, Wolford E. Low rates of headache and migraine associated with intravenous immunoglobulin infusion using a 15-minute rate escalation protocol in 123 patients with primary immunodeficiency. Front Immunol. 2023 Feb 2;13:1075527. doi: 10.3389/fimmu.2022.1075527. eCollection 2022. PMID 36818468
- See also: Sponsor website — http://www.bpl.co.uk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First enrollment: 06 February 2006 Last subject completed: 06 November 2007 Seven investigative sites, all hospital clinics
Pre-assignment Details: This was an open study. All enrolled subjects received study medication.
Groups:
- Gammaplex: All subjects received between 300 to 800 mg/kg/infusion of Gammaplex intravenously, every 21 day or 28 days.
Period: Overall Study
Arm/Group | Gammaplex
Started | 50
Completed | 45
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gammaplex
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 37
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 44.0 (19.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious, Acute, Bacterial Infections (SABIs) Per Subject Per Year in Subjects With Primary Immunodeficiency Disease.
Description: By assessing the number of serious, acute, bacterial infections per subject per year in subjects with Primary Immunodeficiency disease.
Time Frame: 12 months
Population: Intent to Treat (ITT).
Measure: Number; unit: SABIs/subject/year
Arm/Group | Gammaplex
Number analyzed (Participants) | 50
SABIs/subject/year | 0
Statistical Analysis 1: Comparison: Gammaplex; The estimated serious acute bacterial infection (SABI) rate was calculated by dividing no. of infections by no.of subject years. The exponential of the upper limit of the 98% 2-sided Confidence Interval (CI) gave the upper, 1-sided, 99% confidence bound, estimated using Poisson regression. The equivalent upper bound per subject year was obtained by dividing this figure by total subject years; Test type: Superiority or Other; p = 0.01, Poisson regression with log link; SABI per subject per year = 0, 99% CI [0 to 0.101] — Mean SABI rate = 0 per subject per year. 1-sided 99% upper confidence bound could not be calculated

2. Secondary Outcome: The Pharmacokinetic (PK) Half-Life of Immunoglobulin G (IgG)
Description: Blood samples for PK analysis were obtained and analysed at 10 different time points, i.e. -5, 0, 60 minutes (min), 24, 48 hours (hrs), 4, 7, 14, 21 and 28 days, at an infusion visit following 6 months of treatment.
Time Frame: -5, 0, 60 minutes (min), 24, 48 hours (hrs), 4, 7, 14, 21 and 28 days
Population: Only 24 of the 45 evaluable subjects participated in the Pharmacokinetic part of the protocol. No data imputation.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Gammaplex
Number analyzed (Participants) | 24
Days | 41.19 (19.19)

3. Secondary Outcome: The Pharmacokinetic (PK) Clearance of Immunoglobulin G (IgG)
Description: as for outcome 2
Time Frame: -5, 0, 60 min, 24, 48 hrs, 4, 7, 14, 21 and 28 days
Population: Only 24 of the 45 evaluable subjects participated in the Pharmacokinetic part of the protocol. No data imputation.
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Gammaplex
Number analyzed (Participants) | 24
mL/day/kg | 0.585 (0.2508)

4. Secondary Outcome: The Pharmacokinetic (PK) Volume of Distribution (Vz)of Immunoglobulin G (IgG)
Description: as for outcome 2
Time Frame: -5, 0, 60 min, 24, 48 hrs, 4, 7, 14, 21 and 28 days
Population: Only 24 of the 45 evaluable subjects participated in the Pharmacokinetic part of the protocol. No data imputation.
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Gammaplex
Number analyzed (Participants) | 24
dL/kg | 0.297 (0.0539)

5. Secondary Outcome: The Pharmacokinetic (PK) Mean Residence Time (MRT) for Inmuunoglobulin G (IgG)
Description: as for outcome 2
Time Frame: -5, 0, 60 min, 24, 48 hrs, 4, 7, 14, 21 and 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Gammaplex
Number analyzed (Participants) | 50
Days | 56.1 (23.06)

ADVERSE EVENTS:
Time Frame: An event was only included in the analysis of Adverse Events (AEs) if it had an onset date between the first Gammaplex infusion and 30 days after the last Gammaplex infusion, inclusive.
Arm/Group | Gammaplex
Serious Adverse Events (participants affected / at risk) | 6/50
Other Adverse Events (participants affected / at risk) | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gammaplex (N=50)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Basal cell carcinoma, 7 millimeter(mm) lesion on left side of nose, Not related - Resolved
Chest Pain (General disorders) | 1 (1) — Chest pain, Possibly related - Resolved. This SAE occurred in the same subject who experienced Thrombosis and Syncope vasovagal.
Gastroenteritis viral (Infections and infestations) | 1 (1) — Viral gastroenteritis, Not related - Resolved
Pneumonia bacterial (Infections and infestations) | 1 (1) — Bacterial pneumonia, Not related - Resolved Diagnosed prior to first Gammaplex infusion. Treatment for bacterial pneumonia began 4 days before the subject's first infusion in the study.
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Pregnancy, Not related - Resolved
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Moderately differentiated squamous cell carcinoma, Not related - Resolved
Syncope vasovagal (Nervous system disorders) | 1 (1) — Syncopal epsisode, vasovagal in etiology, Not related - Resolved. This Serious Adverse Event (SAE) occurred in the same subject who experienced Thrombosis and Chest pain.
Thrombosis (Vascular disorders) | 1 (1) — Blood clot to left arm, Possibly related - Resolved This SAE occurred in the same subject who also experienced Chest Pain and Syncope vasovagal.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gammaplex (N=50)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (19)
Athralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bronchitis (Infections and infestations) | 6 (7)
Bronchitis acute (Infections and infestations) | 4 (5)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 4 (7)
Conjunctivitis (Eye disorders) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Cystitis (Infections and infestations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 10 (13)
Fatigue (General disorders) | 7 (22)
Gastroenteritis viral (Infections and infestations) | 6 (8)
Headache (Nervous system disorders) | 18 (97)
Hypertension (Vascular disorders) | 3 (10)
Influenza (Infections and infestations) | 3 (4)
Insomnia (Psychiatric disorders) | 3 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Nasopharyngitis (Infections and infestations) | 7 (15)
Nausea (Gastrointestinal disorders) | 9 (12)
Pain (General disorders) | 5 (10)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Pyrexia (General disorders) | 15 (26)
Rash (Skin and subcutaneous tissue disorders) | 5 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Sinus headache (Nervous system disorders) | 3 (4)
Sinusitis (Infections and infestations) | 17 (26)
Upper abdominal pain (Gastrointestinal disorders) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 13 (19)
Urinary tract infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the Study results will be allowed only with prior written approval from Sponsor, said consent not to be unreasonably withheld. At the request of Sponsor, the Institution and/or Investigator shall delete any Confidential Information pertaining to Sponsor's Inventions from any proposed publications prior to submitting or presenting the materials. Any and all publications will give appropriate recognition of any support received from Sponsor.